CLINICAL TRIAL: NCT02848872
Title: Evaluation of Tumor and Blood Immune Biomarkers in Resected Non-small Cell Lung Cancer
Acronym: TOP 1502
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00069742
Record Dates: First submitted 2016-05-26; First posted 2016-07-29 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-05

CONDITIONS: Non-small Cell Lung Carcinoma
Keywords: Tumor-infiltrating lymphocytes (TILs)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Resected NSCLC specimens (excess)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NSCLC patients: Resected patients

SUMMARY:
The hypothesis of this study is that functional tumor infiltrating lymphocyte (TIL) isolation from resected lung cancer specimens is feasible, allowing determination of tumor antigen-specific T cell reactivities. The primary objective of this study is to investigate the feasibility of isolating functional tumor infiltrating lymphocytes s(TILs) to determine tumor antigen-specific T cell re-activities in 30 resected lung tumor specimens. Successful isolation of TILs will be defined as collecting 1x10-6 viable, CD45+ mononuclear cells or greater from tumors containing >/=1 gram of excess tissue. If successful isolation of TILs can be obtained from >/= 66% of resected tumor specimens, the protocol will be considered feasible. The primary exploratory objective is to identify immunologic signatures that predict clinical outcomes from cytotoxic chemotherapy and/or immunotherapy.

DETAILED DESCRIPTION:
Investigating tumor infiltrating lymphocytes in Non-small Cell Lung Cancer (NSCLC) is of clinical importance for multiple reasons. Cellular, antigen, and cytokine profiles associated with favorable clinical outcomes after therapy are currently lacking in lung cancer, and these results may lead to the development of clinically important prognostic and predictive biomarkers. Additionally, by determining the specific cell types and antigen targets of effector cells in the microenvironment, strategies can be devised to alter mechanisms regulating tumor immune tolerance. These data may ultimately enable future, novel combinational approaches of anti-tumor therapies through early phase clinical trials designed to improve clinical outcomes for patients with lung cancer. Finally, by correlating immunologic profiles with clinical outcomes (including pathologic response and progression free survival), signatures can be derived to help predict benefit from cytotoxic chemotherapy for patients receiving these treatments.

This study will plan to enroll a total of 30 patients. This number will consist of a combination of early stage NSCLC patients receiving no neoadjuvant therapy, standard neoadjuvant cytotoxic chemotherapy, or immune checkpoint therapy as well as patients with metastatic disease undergoing tumor resection that have received prior systemic therapy of interest, including but not limited to anti-PD1/PDL agents.

Standard diagnostic and staging work up will be performed, including pathologic/histologic diagnosis of cancer. Patients will receive therapy as deemed appropriate by their treating physician as per standard clinical care or as part of a clinical cancer trial. There is no randomization nor stratification. Patients will not receive any information about the assays/research performed as these are for research purposes only.

Data from patients will be extracted from medical records and images. Data elements that will be extracted include the following: age, sex, tumor histology and stage, chemotherapy regimens and immune-modulating therapy dose and schedule, disease response (outcomes).

Tumor specimen samples will be collected at the time of definitive surgical resection of tumor. After the specimen has been processed for margin status and the frozen section assessment of the specimen is complete, a specimen of excess tumor (at least 1gm) will be released and acquired by the tumor immunology correlative science staff for isolation of tumor infiltrating lymphocytes for purposes of this protocol with any remaining tissue to be processed by the Duke Biorepository staff if the subject has consented to biobanking. For those subjects that decline participation in this biorepository tissue will be processed as outlined above.

Blood will be collected prior to surgery to assess activated CD8+ T cells with specificity against tumor antigens and CD4 and CD8 functional memory.

ELIGIBILITY:
Inclusion Criteria:

* Planned standard of care surgical resection, T > 3 cm or metastatic tumor >1 cm
* Age 18 or older
* Signed written ICF
* If neoadjuvant treatment is received, regimens containing either platinum-based chemotherapy or anti-PD1/PDL1 treatment will be allowed.
* Patients with metastatic disease undergoing tumor resection will be eligible if prior treatment has included systemic therapy of interest, including, but not limited to, anti-PD1/PDL agents.

Exclusion Criteria:

* Prisoners or subjects who are compulsorily detained for treatment of either psychiatric or physical (e.g. infectious) illness are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Clinically suspected or pathologically documented NSCLC patients
  * Planned standard of care surgical resection, T > 3 cm or metastatic tumor >1 cm
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Quantity of functional tumor infiltrating lymphocytes (TILs) to determine tumor antigen-specific T cell re-activities. | At surgery (timepoint variable depending on pre-operative therapy)
  Successful isolation of TILs will be defined as collecting 1x10-6 viable, CD45+ mononuclear cells or greater from tumors containing >/= 1 gm excess tissue in 30 resected lung tumor specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Clarke, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States